CLINICAL TRIAL: NCT03121937
Title: Feasibility of a Technology-Based Treatment Support System
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: No longer able to recruit participants
Sponsor: Northwestern University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Stephen Schueller, Assistant Professor of Preventive Medicine, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU00097492; K08MH102336 (NIH)
Record Dates: First submitted 2017-04-11; First posted 2017-04-20 (Actual); Last update posted 2018-10-10 (Actual); Status verified 2017-04

CONDITIONS: Depression; Depressive Disorder, Major
MeSH Terms: conditions — Depression; Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile App (Experimental): Participants will receive a mobile app to be used during psychotherapy that syncs information with the participant's therapist from sessions.
  Interventions: Behavioral: Mobile App
- Treatment as Usual (No Intervention): Participants will receive treatment as usual with aspects of the mobile app available through paper-based worksheets.

INTERVENTIONS:
Behavioral: Mobile App — The mobile app "mConnect" is an app designed to facilitate psychotherapy for depression and includes mood tracking, goal setting, and communication
  Arms: Mobile App

SUMMARY:
This study aims to evaluate a technology-based treatment support system for patients undergoing the treatment of depression. The investigators will explore the usefulness of the technology-based treatment support system as an adjunct to psychotherapy for depression.

DETAILED DESCRIPTION:
This study aims to evaluate a technology-based treatment support system "mConnect" for patients undergoing the treatment of depression. This system will be evaluated by conducting a randomized controlled trial where patients will either receive the mConnect mobile app or treatment as usual.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* English-speaking
* Currently enrolled in outpatient treatment
* Current diagnosis of major depressive disorder
* Ownership of a smartphone device compatible with the mobile app

Exclusion Criteria

* visual, hearing, voice, or motor impairment that would prevent completion of the study procedures or use of mobile phone
* diagnosis of a psychotic disorder, bipolar disorder, dissociative disorder, substance use disorder, or other diagnosis for which participation in this trial is inappropriate, severe suicidality (has ideation, plan, and intent).
* having completed more than 3 sessions of psychotherapy with current therapist

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Retention | 8 weeks
  Number of completed sessions
Adherence | 8 weeks
  The use of the mobile app. This data will be collected passively by the mobile app sending the following information to the secure server: the date and time the mobile app is launched, the date and time any information is entered into the mobile app, the content of any information entered into the mobile app, the date and time any lessons within the mobile app are read by the participant.
Satisfaction | 8 weeks
  Participant satisfaction with the mobile app will be assessed with a patient version of the Mobile App Rating Scale (MARS) that addresses engagement, functionality, aesthestics, information quality, and one subjective rating of the app as a whole.

SECONDARY OUTCOMES:
Depression | 8 weeks
  Depression as measured by the PHQ-9

CONTACTS AND LOCATIONS:
Overall Officials: Stephen M Schueller, PhD, Principal Investigator — Northwestern University
Locations (1):
- Amita Health, Arlington Heights, Illinois, United States

IPD SHARING:
Plan to Share IPD: No